CLINICAL TRIAL: NCT03813381
Title: The Impact of a Moderate CAlorie and Protein REstriction PROgram (CARE-PRO) as an Efficient and Affordable Therapeutic Strategy in Patients With Barrett's Esophagus.
Brief Title: CAlorie and Protein REstriction PROgram in Barrett's Esophagus Patients (CARE-PRO).
Acronym: CARE-PRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CARE-PRO
Record Dates: First submitted 2019-01-09; First posted 2019-01-23 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Barrett's Esophagus; Overweight and Obesity
Keywords: Esophageal adenocarcinoma; Diet; Physical activity; Microbiota
MeSH Terms: conditions — Barrett Esophagus; Overweight; Obesity; Adenocarcinoma Of Esophagus; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (IA) (Experimental): Patients randomized in the Intervention Arm (IA) will be given personalized diet based on calorie and protein restriction. Calorie restriction will be up to 600 kcal below patients' energy requirements and the amount of protein will be 0.8g of protein/Kg body weight mostly form plant-origin food.
  Interventions: Behavioral: Calorie and protein restriction diet
- Control Arm (CA) (No Intervention): Participants in the CA will be given information about the importance of a healthy lifestyle in reducing the risk of cancer and will receive a leaflet based on WCRF/AICR recommendations.

INTERVENTIONS:
Behavioral: Calorie and protein restriction diet — Patient in intervention arm will be given individualized dietary advice on the basis of WCRF/AICR recommendations. The aim of healthy dietary advice will be the reduction of patient's total daily calorie intake up to 600 kcal below their energy requirements and 0.8g of protein/Kg body weight mostly form plant-origin food.
  Patients, periodically, will meet the dietitian for a 45-minute nutritional counselling session and a trained nurse for a 15-minute health coaching session.
  Each patient in the IA will be involved in at least three 4-hour cooking classes.
  Patients in the IA, after a medical/cardiac evaluation to assure their physical ability for exercise, will attend Nordic walking sessions of moderate intensity two times per month during the 24 months of intervention.
  Arms: Intervention Arm (IA)

SUMMARY:
The increasing incidence of Esophageal Adenocarcinoma (EAC) in several Western countries can be primarily ascribed to risk factors such as obesity, chronic gastroesophageal reflux, dietary habits and alcohol intake. Nevertheless, Barrett's Esophagus (BE), remains the main risk factor for EAC. Several studies supports the role played by the gut microbiota on the modulation of metabolic and immunological pathways. An abnormal state of the microbial ecosystem seems to be involved in the promotion and onset of various diseases, including cancer. Recent studies have shown that diet and lifestyle have an important modulatory role as protective or risk factors for oncological diseases. The World Cancer Research Fund (WCRF) and the American Institute for Cancer Research (AICR) released a review of the evidence that emerged from published studies in the field of nutrition and cancer prevention and summarized their findings into 10 recommendations. Several studies have also shown that a moderate caloric and/or protein restriction seems to be able to reduce the risk of neoplastic disease development. The primary aim of this study is to evaluate the impact of a lifestyle-oriented intervention on body weight, waist circumference, biomarkers associated with cancer risk, esophageal microbiota composition and adherence to cancer prevention recommendations after 24 months in overweight or obese BE patients.

Methods and analysis: Patients are randomly divided into two arms, a control arm (CA) and an interventional arm (IA). The CA receives information about a correct lifestyle to prevent cancer.

The IA is involved in the two-year program of moderate caloric and protein restriction.

At the time of enrollment, anthropometric measurements will be recorded for each patient and they will be randomized to IA or CA. Blood samples will be obtained from each patient and blood glucose will be determined. Serum metabolic biomarkers will be measured in each serum sample and total proteins will be extracted from fresh frozen esophageal biopsy and will be analyzed to evaluate the insulin signal pathway.

To assess esophageal microbiota profiling, total genomic DNA (gDNA) will be extracted from matched fresh frozen biopsy.

In order to determine a score of adherence to cancer prevention recommendations, participants will be asked to complete a self-administrated questionnaire reflecting WCRF/AICR recommendations.

All the measurements will also occur at the end point, after two years from the enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of Barrett's esophagus without dysplasia or cancer aged ≥ 18 years with BMI ≥ 25.0 kg/m^2
* Willingness and ability to perform supervised Nordic walking session twice a month and self-planned physical activity at least 3 times a week
* Signed informed consent

Exclusion Criteria:

* No histological confirmation of Barrett's esophagus
* Cancer diagnosis within one year before trial begins
* Presence of insulin-dependent diabetes
* Denied informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Body weight change | Baseline and after 24 months
  A 7% weight loss

SECONDARY OUTCOMES:
Metabolic serum biomarkers | Baseline and after 24 months
  Fasting glucose (mg/dl)
Metabolic serum biomarkers | Baseline and after 24 months
  Insulin (pg/ml) and C-peptide (pg/ml), tumor necrosis factor-alpha -TNF-alpha (pg/ml) and Interleukin-6 - IL-6 (pg/ml).
Metabolic serum biomarkers | Baseline and after 24 months
  Insulin-like growth factor - IGF1 (nmol/ml), insulin-like growth factor binding protein 1 and 3 - IGFBP1 (nmol/ml) and IGFBP3 (nmol/ml)
Metabolic serum biomarkers | Baseline and after 24 months
  Leptin (ng/ml)
Metabolic serum biomarkers | Baseline and after 24 months
  Adiponectin (µg/ml)
Insulin resistance index (HOMA-IR) | Baseline and after 24 months
  HOMA-IR index [fasting plasma glucose (mg/dl) × fasting serum insulin(μU/ml)/405]
Expression of proteins involved on insulin and IGF1 receptors signal transduction | Baseline and after 24 months
  Phosphoinositide 3-kinases (PI3K)/Protein kinase B(Akt) pathway; mitogenic (ERK/MAPK) pathway
Esophageal microbiota composition | Baseline and after 24 months
  To assess esophageal microbiota profiling, total gDNA will be extracted from fresh frozen biopsy. Specific primers for the bacterial V3-V4 hypervariable regions of 16S ribosomal ribonucleic acid (rRNA) will be used to amplify bacterial DNA [≈ 500 bases pair (bp)] to be sequenced by Illumina Miseq platform with 300 bp paired-end approach.
Adherence score to World Cancer Research Fund and the American Institute for Cancer Research (WCRF/AICR) recommendations for cancer prevention. | Baseline and after 24 months
  In order to determine a score of adherence to cancer prevention recommendations, participants will be asked to complete a 6-item self-administrated questionnaire reflecting six recommendations provided by the World Cancer Research Fund and the American Institute for Cancer Research (WCRF/AICR).
  A score of 1 will be assigned when the item is met and a score of 0 will be assigned when it is not. An answer that partially satisfies the item will be assigned a score of 0.5. Some recommendation (item) have sub-item (item 3,4 and 5). Even for sub-item the score will be 1-0 with 0.5 for partially satisfied item. For total score of item presenting sub-item, we will consider the score obtained by calculating the average score between the sub-item.
  The final adherence score will derive from the mathematical sum of the individual scores obtained for each item. The maximum expected score will be equal to 6 (full adherence).
Waist circumference reduction | Baseline and after 24 months
  Waist circumference (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Realdon, MD, PhD, Principal Investigator — Veneto Institute of Oncology IOV-IRCCS, Padua, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Y Lee C. The Effect of High-Fat Diet-Induced Pathophysiological Changes in the Gut on Obesity: What Should be the Ideal Treatment? Clin Transl Gastroenterol. 2013 Jul 11;4(7):e39. doi: 10.1038/ctg.2013.11. PMID 23842483
- [Background] Teng JA, Wu SG, Chen JX, Li Q, Peng F, Zhu Z, Qin J, He ZY. The Activation of ERK1/2 and JNK MAPK Signaling by Insulin/IGF-1 Is Responsible for the Development of Colon Cancer with Type 2 Diabetes Mellitus. PLoS One. 2016 Feb 22;11(2):e0149822. doi: 10.1371/journal.pone.0149822. eCollection 2016. PMID 26901856
- [Background] Zhu N, Zhang Y, Gong YI, He J, Chen X. Metformin and lung cancer risk of patients with type 2 diabetes mellitus: A meta-analysis. Biomed Rep. 2015 Mar;3(2):235-241. doi: 10.3892/br.2015.417. Epub 2015 Jan 9. PMID 26075077
- [Background] Jemal A, Center MM, DeSantis C, Ward EM. Global patterns of cancer incidence and mortality rates and trends. Cancer Epidemiol Biomarkers Prev. 2010 Aug;19(8):1893-907. doi: 10.1158/1055-9965.EPI-10-0437. Epub 2010 Jul 20. PMID 20647400
- [Background] Vingeliene S, Chan DSM, Vieira AR, Polemiti E, Stevens C, Abar L, Navarro Rosenblatt D, Greenwood DC, Norat T. An update of the WCRF/AICR systematic literature review and meta-analysis on dietary and anthropometric factors and esophageal cancer risk. Ann Oncol. 2017 Oct 1;28(10):2409-2419. doi: 10.1093/annonc/mdx338. PMID 28666313
- [Background] World Cancer Research Fund/American Institute for Cancer Research. Continuous Update Project Report: Diet, Nutrition, Physical Activity and Oesophageal Cancer. 2016. Available at: wcrf.org/oesophageal-cancer-2016. 2016. http://wcrf.org/oesophageal-cancer-2016.
- [Background] De Ceglie A, Fisher DA, Filiberti R, Blanchi S, Conio M. Barrett's esophagus, esophageal and esophagogastric junction adenocarcinomas: the role of diet. Clin Res Hepatol Gastroenterol. 2011 Jan;35(1):7-16. doi: 10.1016/j.gcb.2010.08.015. PMID 20970272
- [Background] Mayne ST, Navarro SA. Diet, obesity and reflux in the etiology of adenocarcinomas of the esophagus and gastric cardia in humans. J Nutr. 2002 Nov;132(11 Suppl):3467S-3470S. doi: 10.1093/jn/132.11.3467S. PMID 12421872
- [Background] Pera M, Manterola C, Vidal O, Grande L. Epidemiology of esophageal adenocarcinoma. J Surg Oncol. 2005 Dec 1;92(3):151-9. doi: 10.1002/jso.20357. PMID 16299786
- [Background] Vaughan TL, Davis S, Kristal A, Thomas DB. Obesity, alcohol, and tobacco as risk factors for cancers of the esophagus and gastric cardia: adenocarcinoma versus squamous cell carcinoma. Cancer Epidemiol Biomarkers Prev. 1995 Mar;4(2):85-92. PMID 7742727
- [Background] Shaheen NJ, Richter JE. Barrett's oesophagus. Lancet. 2009 Mar 7;373(9666):850-61. doi: 10.1016/S0140-6736(09)60487-6. PMID 19269522
- [Background] Cameron AJ, Ott BJ, Payne WS. The incidence of adenocarcinoma in columnar-lined (Barrett's) esophagus. N Engl J Med. 1985 Oct 3;313(14):857-9. doi: 10.1056/NEJM198510033131404. PMID 4033716
- [Background] Bhat S, Coleman HG, Yousef F, Johnston BT, McManus DT, Gavin AT, Murray LJ. Risk of malignant progression in Barrett's esophagus patients: results from a large population-based study. J Natl Cancer Inst. 2011 Jul 6;103(13):1049-57. doi: 10.1093/jnci/djr203. Epub 2011 Jun 16. PMID 21680910
- [Background] Hvid-Jensen F, Pedersen L, Drewes AM, Sorensen HT, Funch-Jensen P. Incidence of adenocarcinoma among patients with Barrett's esophagus. N Engl J Med. 2011 Oct 13;365(15):1375-83. doi: 10.1056/NEJMoa1103042. PMID 21995385
- [Background] Runge TM, Abrams JA, Shaheen NJ. Epidemiology of Barrett's Esophagus and Esophageal Adenocarcinoma. Gastroenterol Clin North Am. 2015 Jun;44(2):203-31. doi: 10.1016/j.gtc.2015.02.001. Epub 2015 Apr 9. PMID 26021191
- [Background] Siegel R, Naishadham D, Jemal A. Cancer statistics, 2013. CA Cancer J Clin. 2013 Jan;63(1):11-30. doi: 10.3322/caac.21166. Epub 2013 Jan 17. PMID 23335087
- [Background] Gordon LG, Mayne GC, Hirst NG, Bright T, Whiteman DC; Australian Cancer Study Clinical Follow-Up Study; Watson DI. Cost-effectiveness of endoscopic surveillance of non-dysplastic Barrett's esophagus. Gastrointest Endosc. 2014 Feb;79(2):242-56.e6. doi: 10.1016/j.gie.2013.07.046. Epub 2013 Sep 27. PMID 24079411
- [Background] Spechler SJ. Barrett esophagus and risk of esophageal cancer: a clinical review. JAMA. 2013 Aug 14;310(6):627-36. doi: 10.1001/jama.2013.226450. PMID 23942681
- [Background] Zhang HY, Spechler SJ, Souza RF. Esophageal adenocarcinoma arising in Barrett esophagus. Cancer Lett. 2009 Mar 18;275(2):170-7. doi: 10.1016/j.canlet.2008.07.006. Epub 2008 Aug 13. PMID 18703277
- [Background] Corley DA, Mehtani K, Quesenberry C, Zhao W, de Boer J, Weiss NS. Impact of endoscopic surveillance on mortality from Barrett's esophagus-associated esophageal adenocarcinomas. Gastroenterology. 2013 Aug;145(2):312-9.e1. doi: 10.1053/j.gastro.2013.05.004. Epub 2013 May 11. PMID 23673354
- [Background] Pohl H, Sirovich B, Welch HG. Esophageal adenocarcinoma incidence: are we reaching the peak? Cancer Epidemiol Biomarkers Prev. 2010 Jun;19(6):1468-70. doi: 10.1158/1055-9965.EPI-10-0012. Epub 2010 May 25. PMID 20501776
- [Background] Ryan AM, Duong M, Healy L, Ryan SA, Parekh N, Reynolds JV, Power DG. Obesity, metabolic syndrome and esophageal adenocarcinoma: epidemiology, etiology and new targets. Cancer Epidemiol. 2011 Aug;35(4):309-19. doi: 10.1016/j.canep.2011.03.001. Epub 2011 Apr 5. PMID 21470937
- [Background] Alberti KG, Zimmet P, Shaw J. Metabolic syndrome--a new world-wide definition. A Consensus Statement from the International Diabetes Federation. Diabet Med. 2006 May;23(5):469-80. doi: 10.1111/j.1464-5491.2006.01858.x. PMID 16681555
- [Background] Cowey S, Hardy RW. The metabolic syndrome: A high-risk state for cancer? Am J Pathol. 2006 Nov;169(5):1505-22. doi: 10.2353/ajpath.2006.051090. PMID 17071576
- [Background] Festa A, D'Agostino R Jr, Williams K, Karter AJ, Mayer-Davis EJ, Tracy RP, Haffner SM. The relation of body fat mass and distribution to markers of chronic inflammation. Int J Obes Relat Metab Disord. 2001 Oct;25(10):1407-15. doi: 10.1038/sj.ijo.0801792. PMID 11673759
- [Background] Tsigos C, Kyrou I, Chala E, Tsapogas P, Stavridis JC, Raptis SA, Katsilambros N. Circulating tumor necrosis factor alpha concentrations are higher in abdominal versus peripheral obesity. Metabolism. 1999 Oct;48(10):1332-5. doi: 10.1016/s0026-0495(99)90277-9. PMID 10535400
- [Background] Aleman JO, Eusebi LH, Ricciardiello L, Patidar K, Sanyal AJ, Holt PR. Mechanisms of obesity-induced gastrointestinal neoplasia. Gastroenterology. 2014 Feb;146(2):357-373. doi: 10.1053/j.gastro.2013.11.051. Epub 2013 Dec 6. PMID 24315827
- [Background] Gallagher EJ, LeRoith D. The proliferating role of insulin and insulin-like growth factors in cancer. Trends Endocrinol Metab. 2010 Oct;21(10):610-8. doi: 10.1016/j.tem.2010.06.007. Epub 2010 Jul 19. PMID 20663687
- [Background] Simone BA, Champ CE, Rosenberg AL, Berger AC, Monti DA, Dicker AP, Simone NL. Selectively starving cancer cells through dietary manipulation: methods and clinical implications. Future Oncol. 2013 Jul;9(7):959-76. doi: 10.2217/fon.13.31. PMID 23837760
- [Background] Arcidiacono D, Dedja A, Giacometti C, Fassan M, Nucci D, Francia S, Fabris F, Zaramella A, Gallagher EJ, Cassaro M, Rugge M, LeRoith D, Alberti A, Realdon S. Hyperinsulinemia Promotes Esophageal Cancer Development in a Surgically-Induced Duodeno-Esophageal Reflux Murine Model. Int J Mol Sci. 2018 Apr 14;19(4):1198. doi: 10.3390/ijms19041198. PMID 29662006
- [Background] Arcidiacono D, Antonello A, Fassan M, Nucci D, Morbin T, Agostini M, Nitti D, Rugge M, Alberti A, Battaglia G, Realdon S. Insulin promotes HER2 signaling activation during Barrett's Esophagus carcinogenesis. Dig Liver Dis. 2017 Jun;49(6):630-638. doi: 10.1016/j.dld.2017.01.154. Epub 2017 Jan 22. PMID 28185837
- [Background] Di Pilato V, Freschi G, Ringressi MN, Pallecchi L, Rossolini GM, Bechi P. The esophageal microbiota in health and disease. Ann N Y Acad Sci. 2016 Oct;1381(1):21-33. doi: 10.1111/nyas.13127. Epub 2016 Jul 14. PMID 27415419
- [Background] Snider EJ, Freedberg DE, Abrams JA. Potential Role of the Microbiome in Barrett's Esophagus and Esophageal Adenocarcinoma. Dig Dis Sci. 2016 Aug;61(8):2217-2225. doi: 10.1007/s10620-016-4155-9. Epub 2016 Apr 11. PMID 27068172
- [Background] Yamashiro Y. Gut Microbiota in Health and Disease. Ann Nutr Metab. 2017;71(3-4):242-246. doi: 10.1159/000481627. Epub 2017 Nov 14. PMID 29136611
- [Background] Gao R, Gao Z, Huang L, Qin H. Gut microbiota and colorectal cancer. Eur J Clin Microbiol Infect Dis. 2017 May;36(5):757-769. doi: 10.1007/s10096-016-2881-8. Epub 2017 Jan 7. PMID 28063002
- [Background] Compare D, G. N. The bacteria-hypothesis of colorectal cancer: pathogenetic and therapeutic implications. Transl Gastrointest Cancer 2013;3:44-53. doi:10.3978/j.issn.2224-4778.2013.05.37
- [Background] Yang L, Lu X, Nossa CW, Francois F, Peek RM, Pei Z. Inflammation and intestinal metaplasia of the distal esophagus are associated with alterations in the microbiome. Gastroenterology. 2009 Aug;137(2):588-97. doi: 10.1053/j.gastro.2009.04.046. Epub 2009 Apr 23. PMID 19394334
- [Background] World Cancer Research Fund/American Institute for Cancer Research, Research AI for C. Food, Nutrition, Physical Activity, and the Prevention of Cancer: a Global Perspective. Washington DC: : American Institute for Cancer Research 2007.
- [Background] Romaguera D, Vergnaud AC, Peeters PH, van Gils CH, Chan DS, Ferrari P, Romieu I, Jenab M, Slimani N, Clavel-Chapelon F, Fagherazzi G, Perquier F, Kaaks R, Teucher B, Boeing H, von Rusten A, Tjonneland A, Olsen A, Dahm CC, Overvad K, Quiros JR, Gonzalez CA, Sanchez MJ, Navarro C, Barricarte A, Dorronsoro M, Khaw KT, Wareham NJ, Crowe FL, Key TJ, Trichopoulou A, Lagiou P, Bamia C, Masala G, Vineis P, Tumino R, Sieri S, Panico S, May AM, Bueno-de-Mesquita HB, Buchner FL, Wirfalt E, Manjer J, Johansson I, Hallmans G, Skeie G, Benjaminsen Borch K, Parr CL, Riboli E, Norat T. Is concordance with World Cancer Research Fund/American Institute for Cancer Research guidelines for cancer prevention related to subsequent risk of cancer? Results from the EPIC study. Am J Clin Nutr. 2012 Jul;96(1):150-63. doi: 10.3945/ajcn.111.031674. Epub 2012 May 16. PMID 22592101
- [Background] Fontana L, Adelaiye RM, Rastelli AL, Miles KM, Ciamporcero E, Longo VD, Nguyen H, Vessella R, Pili R. Dietary protein restriction inhibits tumor growth in human xenograft models. Oncotarget. 2013 Dec;4(12):2451-61. doi: 10.18632/oncotarget.1586. PMID 24353195
- [Background] Fontana L, Partridge L, Longo VD. Extending healthy life span--from yeast to humans. Science. 2010 Apr 16;328(5976):321-6. doi: 10.1126/science.1172539. PMID 20395504
- [Background] Omodei D, Fontana L. Calorie restriction and prevention of age-associated chronic disease. FEBS Lett. 2011 Jun 6;585(11):1537-42. doi: 10.1016/j.febslet.2011.03.015. Epub 2011 Mar 12. PMID 21402069
- [Background] Roberts SB, Speakman J. Update on human calorie restriction research. Adv Nutr. 2013 Sep 1;4(5):563-4. doi: 10.3945/an.113.004317. PMID 24038258
- [Background] Sell Ch. Caloric restriction and insulin-like growth factors in aging and cancer. Horm Metab Res. 2003 Nov-Dec;35(11-12):705-11. doi: 10.1055/s-2004-814156. PMID 14710349
- [Background] Speakman JR, Mitchell SE. Caloric restriction. Mol Aspects Med. 2011 Jun;32(3):159-221. doi: 10.1016/j.mam.2011.07.001. Epub 2011 Aug 10. PMID 21840335
- [Background] Anderson AS, Craigie AM, Caswell S, Treweek S, Stead M, Macleod M, Daly F, Belch J, Rodger J, Kirk A, Ludbrook A, Rauchhaus P, Norwood P, Thompson J, Wardle J, Steele RJ. The impact of a bodyweight and physical activity intervention (BeWEL) initiated through a national colorectal cancer screening programme: randomised controlled trial. BMJ. 2014 Mar 7;348:g1823. doi: 10.1136/bmj.g1823. PMID 24609919
- [Background] Demark-Wahnefried W, Clipp EC, Lipkus IM, Lobach D, Snyder DC, Sloane R, Peterson B, Macri JM, Rock CL, McBride CM, Kraus WE. Main outcomes of the FRESH START trial: a sequentially tailored, diet and exercise mailed print intervention among breast and prostate cancer survivors. J Clin Oncol. 2007 Jul 1;25(19):2709-18. doi: 10.1200/JCO.2007.10.7094. PMID 17602076
- [Background] Admiraal WM, Vlaar EM, Nierkens V, Holleman F, Middelkoop BJ, Stronks K, van Valkengoed IG. Intensive lifestyle intervention in general practice to prevent type 2 diabetes among 18 to 60-year-old South Asians: 1-year effects on the weight status and metabolic profile of participants in a randomized controlled trial. PLoS One. 2013 Jul 22;8(7):e68605. doi: 10.1371/journal.pone.0068605. Print 2013. PMID 23894322
- [Background] Peters NC, Contento IR, Kronenberg F, Coleton M. Adherence in a 1-year whole foods eating pattern intervention with healthy postmenopausal women. Public Health Nutr. 2014 Dec;17(12):2806-15. doi: 10.1017/S1368980014000044. PMID 24499772
- [Background] Villarini A, Pasanisi P, Raimondi M, Gargano G, Bruno E, Morelli D, Evangelista A, Curtosi P, Berrino F. Preventing weight gain during adjuvant chemotherapy for breast cancer: a dietary intervention study. Breast Cancer Res Treat. 2012 Sep;135(2):581-9. doi: 10.1007/s10549-012-2184-4. Epub 2012 Aug 8. PMID 22869285
- [Background] Demark-Wahnefried W, Jones LW. Promoting a healthy lifestyle among cancer survivors. Hematol Oncol Clin North Am. 2008 Apr;22(2):319-42, viii. doi: 10.1016/j.hoc.2008.01.012. PMID 18395153
- [Background] Hawkes AL, Chambers SK, Pakenham KI, Patrao TA, Baade PD, Lynch BM, Aitken JF, Meng X, Courneya KS. Effects of a telephone-delivered multiple health behavior change intervention (CanChange) on health and behavioral outcomes in survivors of colorectal cancer: a randomized controlled trial. J Clin Oncol. 2013 Jun 20;31(18):2313-21. doi: 10.1200/JCO.2012.45.5873. Epub 2013 May 20. PMID 23690410
- [Background] Ligibel JA, Meyerhardt J, Pierce JP, Najita J, Shockro L, Campbell N, Newman VA, Barbier L, Hacker E, Wood M, Marshall J, Paskett E, Shapiro C. Impact of a telephone-based physical activity intervention upon exercise behaviors and fitness in cancer survivors enrolled in a cooperative group setting. Breast Cancer Res Treat. 2012 Feb;132(1):205-13. doi: 10.1007/s10549-011-1882-7. Epub 2011 Nov 24. PMID 22113257
- [Background] Morey MC, Snyder DC, Sloane R, Cohen HJ, Peterson B, Hartman TJ, Miller P, Mitchell DC, Demark-Wahnefried W. Effects of home-based diet and exercise on functional outcomes among older, overweight long-term cancer survivors: RENEW: a randomized controlled trial. JAMA. 2009 May 13;301(18):1883-91. doi: 10.1001/jama.2009.643. PMID 19436015
- [Background] Neuner-Jehle S, Schmid M, Gruninger U. The "Health Coaching" programme: a new patient-centred and visually supported approach for health behaviour change in primary care. BMC Fam Pract. 2013 Jul 17;14:100. doi: 10.1186/1471-2296-14-100. PMID 23865509
- [Background] Pekmezi DW, Demark-Wahnefried W. Updated evidence in support of diet and exercise interventions in cancer survivors. Acta Oncol. 2011 Feb;50(2):167-78. doi: 10.3109/0284186X.2010.529822. Epub 2010 Nov 24. PMID 21091401
- [Background] Vallance JK, Courneya KS, Plotnikoff RC, Yasui Y, Mackey JR. Randomized controlled trial of the effects of print materials and step pedometers on physical activity and quality of life in breast cancer survivors. J Clin Oncol. 2007 Jun 10;25(17):2352-9. doi: 10.1200/JCO.2006.07.9988. PMID 17557948
- [Background] Wahab S, Menon U, Szalacha L. Motivational interviewing and colorectal cancer screening: a peek from the inside out. Patient Educ Couns. 2008 Aug;72(2):210-7. doi: 10.1016/j.pec.2008.03.023. Epub 2008 May 8. PMID 18467066
- [Derived] Arcidiacono D, Zaramella A, Fabris F, Sanchez-Rodriguez R, Nucci D, Fassan M, Nardi M, Benna C, Cristofori C, Morbin T, Pucciarelli S, Fantin A, Realdon S. Insulin/IGF-1 Signaling Is Downregulated in Barrett's Esophagus Patients Undergoing a Moderate Calorie and Protein Restriction Program: A Randomized 2-Year Trial. Nutrients. 2021 Oct 17;13(10):3638. doi: 10.3390/nu13103638. PMID 34684639
- See also: Related Info — http://wcrf.org/oesophageal-cancer-2016

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-11): https://cdn.clinicaltrials.gov/large-docs/81/NCT03813381/Prot_SAP_000.pdf